CLINICAL TRIAL: NCT02412241
Title: Establishing Lymphedema and Fibrosis Measures in Oral Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Jie Deng, Assistant Professor, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VICC SUPP 1529; 1R01DE024982-01 (NIH)
Record Dates: First submitted 2015-04-03; First posted 2015-04-09 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Oral Cavity Cancer; Oropharyngeal Cancer; Lymphedema; Fibrosis
MeSH Terms: conditions — Mouth Neoplasms; Oropharyngeal Neoplasms; Lymphedema; Fibrosis | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LEF Measures (Other): PATIENT-REPORTED OUTCOME MEASURE: Validity of LSIDS-H&N will be assessed using 6 forms (e.g., Vanderbilt Head and Neck Symptom Survey (v2.0); Neck Disability Index; and Hospital Anxiety and Depression Scale).
  CLINICIAN-REPORTED OUTCOME MEASURES: External LEF will be assessed using HN-LEF Grading Criteria, CTCAE (v4.03), and digital photos of the head and neck. Internal LEF will be scored using Modified Patterson Scale through an endoscopic exam. Both external/internal measures are re-assessed for intrarater and interrater reliability.
  OBJECTIVE/TECHNICAL MEASURES: Patients undergo CT scans and ultrasound exams with results re-scored for intrarater and interrater reliability.
  Interventions: Other: LEF measures; Procedure: Technical measure

INTERVENTIONS:
Other: LEF measures — Patient-reported outcome measure; clinician-reported outcome measures
Procedure: Technical measure — Undergo standard CT scan
  Other Names: Computed Tomography (CT)
Procedure: Technical measure — Undergo standard ultrasound
  Other Names: Ultrasonography, Ultrasound (US) Medical Ultrasound

SUMMARY:
This four-year, prospective, longitudinal study will evaluate and validate a patient-reported outcome measure, clinician-reported outcome measures, and imaging techniques in assessing characteristics, trajectory, and progression of lymphedema and fibrosis (LEF) in oral cavity and oropharyngeal cancer patients.

This clinical trial studies patient-and-clinician-reported measures as well as standard imaging methods to see how accurate they are in identifying and evaluating lymphedema (swelling) or fibrosis (tough or tight tissue) in the head and neck region of patients receiving treatment for newly diagnosed stage II-IV oral cavity or oropharyngeal cancer. Lymphedema and fibrosis (LEF) can lead to physical symptoms, such as trouble swallowing and chewing, as well as psychological and emotional symptoms, such as negative body image and avoiding social interactions. Finding an accurate test to identify and evaluate LEF may allow doctors to treat LEF more quickly and control symptoms more effectively, and thus provide patients with a better quality of life.

DETAILED DESCRIPTION:
The goal of this proposed study is to establish a valid, clinically useful measurement battery for head and neck LEF by achieving these specific aims:

Aim 1: To determine the reliability and validity of the patient-reported outcome measure (LSIDS-H&N) for assessing LEF-related symptoms in oral cavity and oropharyngeal cancer patients across the trajectory of treatment, recovery, and survival.

Aim 2: To determine the reliability and validity of the clinician-reported outcome measures (HN-LEF Grading Criteria and Modified Patterson Scale) for assessing external and internal LEF in oral cavity and oropharyngeal cancer patients across the trajectory of treatment, recovery, and survival.

Aim 3: To determine the reliability and validity of imaging techniques (CT scan and ultrasonography) in identifying site-specific LEF in oral cavity and oropharyngeal cancer patients across the trajectory of treatment, recovery, and survival.

ELIGIBILITY:
Inclusion Criteria:

* a newly diagnosed, histologically proven cancer arising from the oral cavity and oropharynx
* tumor stage II or greater
* age ≥ 21 years old
* willing and able to undergo study assessment
* able to speak and read English and understand Informed Consent.

Exclusion Criteria:

* have medical record documentation of cognitive impairment that would preclude the ability to provide informed consent
* are unwilling to undergo routine follow-up
* have recurrent cancer
* have any other active cancer.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2015-06; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Reliability of the patient-reported outcome measure (LSIDS-H&N) in terms of internal consistency of each symptom cluster | Up to 12 months after treatment
  The assessment will be conducted at pre-treatment, end of treatment (EOT), and every three months up to 12 months after treatment

SECONDARY OUTCOMES:
Validity of the patient-reported outcome measure (LSIDS-H&N) in terms of content, construct, sensitivity to change, and clinical feasibility | Up to 12 months after treatment
  The assessment will be conducted at pre-treatment, EOT, and every three months up to 12 months after treatment
Reliability of the clinician-reported outcome measures (HN-LEF Grading criteria and the Modified Patterson Scale) | 12 months after treatment
  The assessment will be conducted at pre-treatment, EOT, and every three months up to 12 months after treatment
Validity of the clinician-reported outcome measures (HN-LEF Grading criteria and the Modified Patterson Scale) in terms of criteria correlations, sensitivity to change, and clinical feasibility | 12 months after treatment
  The assessment will be conducted at pre-treatment, EOT, and every three months up to 12 months after treatment
Reliability of imaging techniques in identifying site-specific LEF across the trajectory of treatment, recovery, and survival | 12 months after treatment
  The assessment will be conducted at pre-treatment, and every three months up to 12 months after treatment
Validity of imaging techniques in identifying site-specific LEF across the trajectory of treatment, recovery, and survival, in terms of concordance correlation, sensitivity to change, and clinical feasibility | 12 months after treatment
  The assessment will be conducted at pre-treatment, and every three months up to 12 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jie Deng, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Vanderbilt Ingram Cancer Center, Find a Clinical Trial — http://vicc.org/ct/